CLINICAL TRIAL: NCT02311413
Title: The Effect of Peptide Immunotherapy on Frequency, Memory Phenotype, Chemokine Receptor Expression and Markers of Regulatory T Cell Function Among Allergen-Specific T Cells
Brief Title: A Randomized Prospective Clinical Trial of Fel d 1 Peptide Immunotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Circassia Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT U19-MMU-02; U19AI100266 (NIH)
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Cat Allergy; Cat Hypersensitivity
Keywords: Allergic rhinoconjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cat-PAD (Experimental): Subjects will be treated with four monthly doses of Cat-PAD, a peptide immunotherapy product consisting of Fel d 1 synthetic peptide immunoregulatory epitopes (SPIRE).
  Interventions: Drug: Cat-PAD
- Placebo (Placebo Comparator): Subjects will be treated with 4 monthly doses of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cat-PAD — The assigned study intervention will be administered by intradermal injection into the flexor surface of the forearm.
  Other Names: ToleroMune Cat
  Arms: Cat-PAD
Drug: Placebo — The assigned study intervention will be administered by intradermal injection into the flexor surface of the forearm.
  Other Names: Cat-PAD Placebo
  Arms: Placebo

SUMMARY:
The goal of this study is to identify changes in cells that are related to the treatment with Cat-PAD (ToleroMune Cat).

DETAILED DESCRIPTION:
Cat-PAD is an experimental cat allergy vaccine and has been studied to determine if it can reduce symptom scores of participants exposed to cat allergen. To study how the vaccine causes changes in the immune system, the researchers plan to evaluate changes in the blood (genes and proteins) and urine in response to the Cat-PAD vaccine.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

* Subject must be able to understand and provide informed consent;
* Subjects without asthma or with asthma who are on Global Initiative for Asthma (GINA) Step 1 treatment with an inhaled short-acting beta2-agonist or GINA Step 2 or 3 treatment with an inhaled corticosteroid. Treatment for asthma must have been stable (drug(s), dose, frequency) for at least 4 weeks prior to randomization. The dose of inhaled corticosteroids must not be greater than 500 microg fluticasone or equivalent (e.g.>00 microg budesonide; or >400 microg mometasone) per day for the treatment of asthma;
* A minimum 1-year documented history of allergic rhinoconjunctivitis on exposure to cats;
* Positive skin prick test to cat hair (wheal diameter 3mm larger than negative control. Cat specific IgE greater than or equal to 0.35IU/ml;
* Subjects must express one (or more) of the following Human Leukocyte Antigens (HLA): HLA-DRB1*0101, HLA-DRB1*0301, HLA-DRB1*0401, HLA-DRB1*0405, HLA- DRB1*0701, HLA-DRB1*0901, HLA-DRB1*1001, HLA-DRB1*1101, HLA-DRB1*1301, HLA-DRB1*1401, HLA-DRB5*0101. Not limited to the above listed HLA as more may become available in the future;
* FEV1 must not decrease >20% from baseline prior to nasal allergen challenges, that does not return to baseline after inhalation of 200µg of Salbutamol. Baseline is defined as the FEV1 value at Visit Pre-Screening;
* Screening nasal allergen challenge in which TNSS is less than or equal to 4 at baseline and greater than or equal to after the highest dose, and

  --Between the first non-zero dose and 10 minutes after the highest dose, either;
  * 3 or more sneezes are counted, or
  * greater than 20% drop in PNIF is recorded, at the discretion of the Physician;
* Subjects must have regular exposure (minimum 1 hour exposure twice per week) to a cat in their normal living or working circumstances;
* Willing and able to comply with the study requirements;
* If the subject is female and of childbearing potential she must have been stable on highly effective contraceptive methods for at least 3 months prior to screening and continue during the study, and produce a negative urine pregnancy test at all visits. Subject may be included without a negative urine pregnancy test if she can document that she is surgically sterile or at least 2 years post-menopausal. Highly effective contraceptive methods may include:

  * Total sexual abstinence for the total duration of the study including washout periods;
  * Vasectomised sexual partner (with appropriate post-vasectomy documentation of the absence of sperm in ejaculate) + male condom;
  * Tubal occlusion + male condom;
  * Intrauterine device (IUD), provided coils are copper banded + male condom;
  * Intrauterine system (IUS) Levonorgestrel, e.g. Mirena + male condom;
  * Medroxyprogesterone injections (Depo-Provera) + male condom;
  * Etonogestrel implants (e.g. Implanon, Norplant) + male condom;
  * Normal and low dose combined oral pills + male condom;
  * Norelgestromin /EE transdermal system + male condom;
  * Intravaginal device, e.g. EE and etonogestrel + male condom;
  * Cerazette(TM) (desogestrel) + male condom.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol;
* Asthma symptoms that have been unstable in the 12 weeks prior to study entry or requirement of oral corticosteroids to treat asthma in the 6 months prior to study entry in the 12 weeks prior to randomization;
* Any history of intubation/life-threatening episode for asthma exacerbation;
* Hospitalization for asthma in the year prior to screening.;
* A history of anaphylaxis to cat allergen. As defined by; (1) more than one organ system involvement with symptoms such as urticaria, wheezing, shortness of breath, abdominal pain, vomiting, (2) presence of hypotension or cyanosis, or loss of consciousness;
* Subjects with an FEV1 <0% of predicted;
* Subjects with an FEV1/FVC ratio of < 70;
* History of significant recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment;
* At time of screening, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Subjects may be re- evaluated for eligibility after symptoms resolve and will maintain the same Subject Screening number;
* The subject has unacceptable symptoms in the 5 days without oral antihistamines prior to the screening visits;
* Treatment with omalizumab within 6 months of screening;
* Previous allergen immunotherapy for cat allergy;
* Subjects for whom administration of epinephrine is contra-indicated;
* Subjects treated with beta-blockers;
* Symptoms of a clinically relevant illness, in the Investigator's opinion, within 6 weeks prior to Screening Visit;
* Female subjects who are pregnant, lactating or planning a pregnancy;
* Any clinically relevant abnormalities on physical examination;
* Vital signs (blood pressure, pulse, respiratory rate, body temperature) outside normal limits unless considered not to be clinically relevant by the Investigator;
* Laboratory values (haematology, biochemistry, urine tests) outside the normal ranges, unless considered not to be clinically relevance by the Investigator. Hemoglobin must be greater than 12g/dl at visits 1, 3 and 4. If the hemoglobin is <12g/dl the visit can be rescheduled within 2 weeks at the discretion of the investigator/physician and the hemoglobin measurement repeated at the subsequent visit;
* History of alcohol or drug abuse;
* History of immunopathological diseases which may confound study outcomes;
* Previous participation in any Cat-PAD study;
* A history of severe drug allergy, severe angioedema or anaphylactic reaction to food;
* Received treatment with an investigational drug within 3 months prior to study;
* Unable to communicate or to understand the requirements of the study, which would impair communication between subject and Investigator thereby interfering with the informed consent procedure or the gathering of study data;
* A history of any significant disease or disorder (e.g. autoimmune, cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, musculoskeletal, endocrine, metabolic, neoplastic/malignant, psychiatric, major physical impairment, severe atopic dermatitis) which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results of the study, or the subject's ability to participate in the study;
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study;
* A known allergy to thioglycerol;
* Known history of positive test results for Hepatitis B, Hepatitis C, HIV or tuberculosis other than would be anticipated following vaccination.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Change in the area under the curve (AUC) from 0 to 6 hour for total nasal symptom score (TNSS). | Following nasal allergen challenge , one year after initiation of peptide immunotherapy.
  This outcome will be analyzed using analysis of covariance (ANCOVA) where the difference in mean AUC between the untreated and treated groups will be compared while statistically controlling for the effects of the baseline AUC.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Neighbour, Principal Investigator — Saint Joseph's Healthcare
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait